CLINICAL TRIAL: NCT02221102
Title: Treatment of Edoxaban Versus Aspirin for Non-disabling Cerebrovascular Events: Rationale, Objectives, and Design
Brief Title: Edoxaban for TIA and Acute Minor Stroke
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Xijing Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Xijing-Edoxaban
Record Dates: First submitted 2014-08-18; First posted 2014-08-20 (Estimated); Last update posted 2014-08-20 (Estimated); Status verified 2014-08

CONDITIONS: Ischemia; Stroke; Cerebral Infarction
Keywords: edoxaban; aspirin; new oral anticoagulant; TIA; acute minor ischemic stroke
MeSH Terms: conditions — Ischemia; Stroke; Cerebral Infarction | interventions — Aspirin; edoxaban

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- aspirin (Active Comparator): Receiving a 100-mg dose of aspirin and placebo edoxaban from day 1 to day 30
  Interventions: Drug: Aspirin; Drug: placebo
- edoxaban 30mg (Experimental): Receiving a 30-mg dose of edoxaban and placebo aspirin from day 1 to day 30
  Interventions: Drug: edoxaban; Drug: placebo
- edoxaban 60mg (Experimental): Receiving a 60-mg dose of edoxaban and placebo aspirin from day 1 to day 30
  Interventions: Drug: edoxaban; Drug: placebo

INTERVENTIONS:
Drug: Aspirin — non-steroidal anti-inflammatory drugs
  Other Names: Acetylsalicylic acid
  Arms: aspirin
Drug: edoxaban — orally active direct factor Xa inhibitor
  Other Names: DU176b; LIXIANA TABLETS
  Arms: edoxaban 30mg; edoxaban 60mg
Drug: placebo

SUMMARY:
Transient ischemic attack (TIA) or minor ischemic stroke has a high risk of early recurrent stroke. As the golden standard, aspirin effect modestly on acute ischemic stroke, and slightly increase the risk of intracerebral hemorrhage. Recently, edoxaban, a new oral anticoagulant, is proved to be as effective as traditional anticoagulants, while carrying significantly less risk of intracranial hemorrhage.

This trial is a randomized, double-blind, multicenter, controlled clinical trial in China. The investigators will assess the hypothesis that a 30-days edoxaban regimen is superior to aspirin alone for the treatment of high-risk patients with acute nondisabling cerebrovascular event.

ELIGIBILITY:
Inclusion Criteria:

* Adult subjects (male or female ≥18 years old)
* Acute nondisabling ischemic stroke (NIHSS ≤3 at the time of randomization) that can be treated with study drug within 24 hours of symptoms onset. Symptom onset is defined by the "last see normal" principle
* TIA (neurologic deficit attributed to focal brain ischemia, with resolution of the deficit within 24 hours of symptom onset), that can be treated with investigational medication within 24 hours of symptoms onset. Symptom onset is defined by the "last see normal" principle
* Informed consent signed

Exclusion Criteria:

* Diagnosis of hemorrhage or other pathology, such as vascular malformation, tumor, abscess or other major nonischemic brain disease, on baseline head CT or MRI scan
* mRS score >2 at randomization (premorbid historical assessment)
* NIHSS ≥4 at randomization
* Clear indication for anticoagulation (atrial fibrillation, mechanical cardiac valves, deep venous thrombosis, pulmonary embolism or known hypercoagulable state)
* Contraindication to investigational medications
* Thrombolysis for ischemic stroke within preceding 7 days
* History of intracranial hemorrhage
* Current treatment (last dose given within 10 days before randomization) with heparin therapy or oral anticoagulation
* Gastrointestinal bleed or major surgery within 3 months
* Planned or likely revascularization (any angioplasty or vascular surgery) within the next 3 months
* TIA or minor stroke induced by angiography or surgery
* Severe noncardiovascular comorbidity with life expectancy <3 months
* Women of childbearing age not practicing reliable contraception who do not have a documented negative pregnancy test result
* Severe renal failure, defined as Glomerular Filtration Rate (GFR) <30 ml/min -Severe hepatic insufficiency (Child-Pugh score B to C)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3700 (Estimated)
Dates: Start 2013-12; Primary Completion 2015-06 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
percentage of patients with new stroke (ischemic or hemorrhage) | 90 days

SECONDARY OUTCOMES:
Percentage of patients with new clinical vascular events (ischemic stroke/hemorrhagic stroke/TIA/myocardial infarction/vascular death) | 30 days
mRS score changes (continuous) and dichotomized at percentage with score 0 to 2 versus 3 to 6 | 30 days and 90 days
Changes in NIHSS scores | 90 days
moderate to severe bleeding events | 90 days
Total mortality | 90 days
Adverse events/severe adverse events reported by the investigators | 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Gang Zhao, M.D., Study Chair — Xijing hostipal
Locations (1):
- Xijing Hospital, Xi'an, Shaanxi, China